CLINICAL TRIAL: NCT00490971
Title: A Randomized, Double-Blind, Active- and Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Extended-Release Paliperidone as Maintenance Treatment After an Acute Manic or Mixed Episode Associated With Bipolar I Disorder
Brief Title: A Study to Evaluate the Effectiveness and Safety of Extended-Release (ER) Paliperidone Compared With Placebo in Delaying the Recurrence of Symptoms in Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR010825; R076477BIM3004 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2007-06-18; First posted 2007-06-25 (Estimated); Results first posted 2012-03-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Mania; Depression; Manic-Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Mania; Depression | interventions — Olanzapine; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paliperidone ER (Experimental)
  Interventions: Drug: Paliperidone ER
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Once daily in dose range of 5 to 20 mg/day for 15 weeks, then until recurrence
  Arms: Olanzapine
Drug: Paliperidone ER — Once daily in dose range of 3 to 12 mg/day for 15 weeks, then until recurrence
  Arms: Paliperidone ER
Drug: Placebo — Once daily until recurrence (only after initial 15 weeks on paliperidone ER)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of oral extended-release (ER) paliperidone compared with placebo in the prevention of the recurrence of mood symptoms in patients with Bipolar I Disorder who initially respond to treatment of an acute manic or mixed episode with paliperidone ER. Olanzapine was included as an active control arm, although the study is not designed to allow for a direct comparison of olanzapine with paliperidone.

DETAILED DESCRIPTION:
This is a randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken), active- and placebo-controlled, parallel-group, multicenter study to evaluate the efficacy (effectiveness) and safety of paliperidone ER relative to placebo in the prevention of recurrent mood symptoms associated with Bipolar I Disorder.

There are 5 phases in this study: a screening phase (lasting up to 7 days) to establish a subject's eligibility for the study,; a 3-week double-blind acute treatment phase to treat the acute or manic episode; a 12-week double-blind treatment continuation phase to establish a patient's clinical stability,; a double-blind treatment maintenance phase to measure the time to symptom recurrence that will last until the patient experiences a recurrence,; and a follow-up phase consisting of a visit approximately 1 week after the last study visit. All antipsychotic drugs and all mood stabilizers other than study drug must be discontinued before the first study drug administration.

Hospitalization is required for at least the first 7 days of the acute treatment phase. At the beginning of the acute treatment phase, patients will be randomly assigned to receive ER paliperidone or olanzapine in a 4:1 ratio. Patients in the ER paliperidone group who have a clinical response at the end of the acute treatment phase, remain clinically stable throughout the continuation phase, and achieve remission for each of the last 3 weeks of the continuation phase will again be randomly assigned: they will be assigned in a 1:1 ratio to receive ER paliperidone or placebo in the maintenance phase. Patients in the olanzapine treatment group who fulfill the same criteria will continue receiving double-blind treatment with olanzapine in the maintenance phase.

Measures of efficacy used are the Young Mania Rating Scale (YMRS), Montgomery-Åsberg Depression Rating Scale (MADRS), Clinical Global Impression - Bipolar Disorder - Severity of Illness Scale (CGI-BP-S), Global Assessment of Functioning (GAF), the Short Form-36 to measure health-related functional status, and the sleep visual analog scale (VAS).

Safety evaluations include monitoring of adverse events, clinical laboratory tests (including urine pregnancy testing and hemoglobin A1c), 12-lead ECG, vital signs measurements, measurement of orthostatic changes in pulse and blood pressure, physical examinations (including height, body weight, and waist circumference), and monitoring of extrapyramidal symptoms using the Abnormal Involuntary Movement Scale (AIMS), the Barnes Akathisia Rating Scale (BARS), and the Simpson Angus Scale (SAS). In addition, the Scale for Suicidal Ideation will be administered to assess suicidality.

The primary hypothesis for this study is that, during the long-term treatment of patients with Bipolar I Disorder who maintain clinical stability after an acute manic or mixed episode, ER paliperidone is superior to placebo in delaying the time to recurrence of any mood symptoms associated with Bipolar I Disorder. Patients begin the acute treatment phase at 6.0 mg/day of oral ER paliperidone or 10 mg/day of oral olanzapine. Dosages may be adjusted, as needed, between 3 to 12 mg/day of ER paliperidone or 5 to 20 mg/day of olanzapine, through the end of the continuation phase. Then, in the maintenance phase, patients receive the dosage of ER paliperidone (or ER paliperidone placebo) or olanzapine reached at the end of the continuation phase. They remain on those dosages until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition) criteria for Bipolar I Disorder Most Recent Episode Manic or Mixed (with or without psychotic features)
* have a history of at least 2 previously documented mood episodes associated with Bipolar I Disorder (1 of which must be a manic or mixed episode) that required medical treatment within the past 3 years
* a total score of at least 20 on the YMRS at screening and at Day 1 of the study.

Exclusion Criteria:

* Meet DSM-IV criteria for any type of episode associated with bipolar disorder other than Bipolar I Disorder Most Recent Episode Manic or Mixed
* Meet DSM-IV criteria for rapid cycling
* Meet DSM-IV criteria for schizoaffective disorder
* Known or suspected borderline or antisocial personality disorder
* be, in the opinion of the investigator, at significant immediate risk for suicidal or violent behavior during the course of the study based on current status or prior history (e.g., suicide attempts during previous episodes).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2006-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (78):
- United States (16):
  - Scottsdale, Arizona
  - Riverside, California
  - San Diego, California
  - Jacksonville, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Willingboro, New Jersey
  - Cincinnati, Ohio
  - Lyndhurst, Ohio
  - Philadelphia, Pennsylvania
  - Arlington, Texas
  - Austin, Texas
  - Bellevue, Washington
- Bulgaria (3):
  - Bulgaria
  - Radnevo
  - Sofia
- China (7):
  - Baoding
  - Beijing
  - Guangzhou
  - Nanjing
  - Shanghai
  - Suzhou
  - Xi'an
- San José, Costa Rica
- France (2):
  - Casablanca
  - Manouba
- Germany (7):
  - Berlin
  - Bochum
  - Chemnitz
  - Düsseldorf
  - Göttingen
  - Jena
  - Lübeck
- India (7):
  - Bangalore
  - Calicut
  - Coimbatore
  - Hyderabad
  - Ludhiana
  - Pune
  - Varanasi
- Kuala Lumpur, Malaysia
- Panama (2):
  - Panama City
  - Panama Panama
- Poland (7):
  - Gdansk
  - Krakow
  - Leszno
  - Skąpe
  - Swiecie Poland
  - Torun
  - Tuszyn
- Romania (5):
  - Bucharest
  - Craiova
  - Iași
  - Tg Mures
  - Timișoara
- Russia (5):
  - Krasnodar
  - Nizny Novgorod
  - Perm
  - Smolensk Region N/A
  - Yaroslavl
- Serbia (4):
  - Belgrade
  - Gornja Toponica
  - Kragujevac
  - Novi Kneževac
- South Africa (4):
  - Cape Town
  - Durban Kn
  - Johannesburg
  - Pretoria
- Turkey (Türkiye) (2):
  - Ankara
  - Manisa
- Ukraine (5):
  - Dnipro
  - Donetsk
  - Kiev
  - Lviv
  - Vinnitsa

REFERENCES:
- [Derived] Berwaerts J, Melkote R, Nuamah I, Lim P. A randomized, placebo- and active-controlled study of paliperidone extended-release as maintenance treatment in patients with bipolar I disorder after an acute manic or mixed episode. J Affect Disord. 2012 May;138(3):247-58. doi: 10.1016/j.jad.2012.01.047. Epub 2012 Feb 27. PMID 22377512

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The double-blind (ie, niether physician nor patient knows the treatment that the patient receives) study has 15-week acute/continuation phase followed by variable-duration maintenance phase (lasting until patient had recurrence or discontinued treatment) to assess effect of paliperidone on maintenance of remission of Bipolar I Disorder
Groups:
- Paliperidone Extented Release (ER): Acute and continuation period. Paliperidone ER: Oral tablet, 3 mg/day to 12 mg/day, Once daily.
- Olanzapine: Acute and continuation period. Olanzapine: Oral tablet, 5 mg/day to 20 mg/day, Once daily.
- Pali/Placebo: Maintenance period. Placebo (Paliperidone in the acute and continuation period).
- Pali/Pali: Maintenance period. Paliperidone ER: Oral tablet, 3 mg/day to 12 mg/day, Once daily (Paliperidone in the acute and continuation period)
- Olan/Olan: Maintenance period. Olanzapine Oral tablet, 5 mg/day to 20 mg/day, Once daily (Olanzapine in the acute and continuation period)
Period: Acute/Continuation
Arm/Group | Paliperidone Extented Release (ER) | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Started | 614 (617 participants were assigned to paliperidone, out of which 614 took the study medication.) | 148 (149 participants were assigned to paliperidone, out of which 148 took the study medication.) | 0 ("0" indicates this group is not relevant to acute and continuation period.) | 0 ("0" indicates this group is not relevant to acute and continuation period.) | 0 ("0" indicates this group is not relevant to acute and continuation period.)
Completed | 308 | 86 | 0 ("0" indicates this group is not relevant to acute and continuation period.) | 0 ("0" indicates this group is not relevant to acute and continuation period.) | 0 ("0" indicates this group is not relevant to acute and continuation period.)
Not Completed | 306 | 62 | 0 | 0 | 0
Not completed — Adverse Event | 62 | 13 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 106 | 12 | 0 | 0 | 0
Not completed — Lost to Follow-up | 23 | 7 | 0 | 0 | 0
Not completed — Protocol Violation | 10 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 92 | 24 | 0 | 0 | 0
Not completed — Other | 11 | 4 | 0 | 0 | 0
Period: Maintenance
Arm/Group | Paliperidone Extented Release (ER) | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Started | 0 ("0" indicates this group is not relevant to maintenance period.) | 0 ("0" indicates this group is not relevant to maintenance period.) | 147 (148 participants were assigned to pali/placebo, out of which 147 took the study medication.) | 149 (152 participants were assigned to pali/pali, out of which 149 took the study medication.) | 83
Completed | 0 ("0" indicates this group is not relevant to maintenance period.) | 0 ("0" indicates this group is not relevant to maintenance period.) | 96 | 96 | 44
Not Completed | 0 | 0 | 51 | 53 | 39
Not completed — Adverse Event | 0 | 0 | 4 | 5 | 7
Not completed — Death | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 5 | 8 | 10
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 4 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 26 | 28 | 18
Not completed — Other | 0 | 0 | 11 | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone ER: Acute and continuation period. Paliperidone ER: Oral tablet, 3 mg/day to 12 mg/day, Once daily.
- Total: Total of all reporting groups
Arm/Group | Paliperidone ER | Olanzapine | Total
Number analyzed (Participants) | 614 | 148 | 762
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 10
  Between 18 and 65 years | 606 | 145 | 751
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (11.93) | 39.2 (11.49) | 39.6 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310 | 80 | 390
  Male | 304 | 68 | 372
Region of Enrollment [Number; unit: participants]
  Asia | 162 | 36 | 198
  Eastern Europe | 129 | 31 | 160
  European Union | 71 | 19 | 90
  North America | 177 | 41 | 218
  Other | 75 | 21 | 96
  India | 69 | 14 | 83
  Malaysia | 7 | 2 | 9
  China | 86 | 20 | 106
  Russian Federation | 51 | 11 | 62
  Serbia | 32 | 8 | 40
  Ukraine | 46 | 12 | 58
  Bulgaria | 27 | 6 | 33
  Germany | 6 | 3 | 9
  Poland | 16 | 5 | 21
  Romania | 22 | 5 | 27
  Costa Rica | 12 | 4 | 16
  Morocco | 6 | 2 | 8
  Panama | 3 | 1 | 4
  South Africa | 26 | 6 | 32
  Tunisia | 10 | 4 | 14
  Turkey | 18 | 4 | 22
  United States | 177 | 41 | 218
AgeCategorical [Number; unit: participants]
  18-25 | 98 | 25 | 123
  26-50 | 378 | 96 | 474
  51-65 | 138 | 27 | 165
  >65 | 0 | 0 | 0
  <18 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence of Any Mood Symptoms (Manic or Depressive) Associated With Bipolar I Disorder
Description: Time to first recurrence of any mood symptoms (ie, manic or depressive) associated with bipolar I disorder during the maintenance phase, after maintaining clinical stability during continued treatment with paliperidone ER over a period of 15 weeks. The time period was from occurrence of acute manic or mixed episode to Week 15. This outcome was measured using combination of various scales, hospitalization for any mood symptoms, use of any medicines for an mood episode and clinical events suggestive of recurrent mood episode associated with bipolar I disorder.
Time Frame: Date of randomization into the maintenance phase until the first occurrence of recurrence of any symptoms or discontinuation from the study, assessed over a period of 41 months.
Population: Intent-to-treat analysis set (ITT) in maintenance (MA) phase, which included participants who entered the MA phase and took at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Number analyzed (Participants) | 0 | 0 | 144 | 146 | 82
Days
  25% Quantile of Time to Recurrence |  |  | 85.0 [72.0 to 141.0] | 140.0 [72.0 to 274.0] | 541 [386.0 to NA] — There were 23% of the subjects in Olan/Olan treatment group who reported recurrence. Hence 25% quantile of time to recurrence was not observed
  Median Time to Recurrence |  |  | 283.0 [203.0 to 531.0] | 558.0 [401.0 to 804.0] | NA [NA to NA] — There were 23% of the subjects in Olan/Olan treatment group who reported recurrence. Hence median time to recurrence was not observed
Statistical Analysis 1: Comparison: Pali/Placebo; Null hypothesis: there is no difference between Pali/Pali and Pali/Placebo in the time to recurrence of any mood symptoms related to bipolar I disorder. An interim analysis was performed when approximately 85% of the required number of recurrences were reported in Pali/Pali and Pali/Placebo treatment groups. A flexible group-sequential approach was adopted. The general family of alpha spending function based on the rho-family with rho=2.5 at overall type I error of 0.025 (1-sided) was employed; Test type: Superiority or Other; p = 0.017, Weighted Z- test — The two treatment groups were compared using a weighted z-statistic based on rho-family of alpha spending function at information fraction of 85.0% at interim analysis analysis (rho=2.5) at 0.025 (1-sided) level. One-sided alpha at final was 0.0195

2. Secondary Outcome: Time to Recurrence of Manic Symptoms Associated With Bipolar I Disorder
Description: This was the key secondary efficacy end-point. Pali/Pali and Pali/Placebo were compared with each other with respect to time to recurrence of manic symptoms. The criterias used for this analysis were similar to criterias used for primary analysis.
Time Frame: Date of randomization into the maintenance phase until the first occurrence of recurrence of manic symptoms or discontinuation from the study, assessed over a period of 41 months.
Population: Intent-to-treat analysis set in MA phase, which included participants who entered the MA phase and took at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Number analyzed (Participants) | 0 | 0 | 144 | 146 | 82
Days
  25% Quantile of Time to Recurrence |  |  | 194.0 [125.0 to 283.0] | 498.0 [294.0 to 813.0] | NA [595.0 to NA] — There were 11% of the subjects in the Olan/Olan group who reported recurrence of manic symptoms. Hence 25% quartile of time to recurrence was not observed.
  Median Time to Recurrence |  |  | 550.0 [419.0 to 878] | NA [813 to NA] — There were 21% of the subjects in the Pali/Pali group who reported recurrence of manic symptoms. Hence median time to recurrence was not observed. | NA [NA to NA] — There were 11% of the subjects in the Olan/Olan group who reported recurrence of manic symptoms. Hence median time to recurrence was not observed.
Statistical Analysis 1: Comparison: Pali/Placebo; At the time of interim analysis of the primary efficacy endpoint, the proportion of recurrence of manic symptoms was 81.9% of the number of recurrence of manic symptoms at final analysis. A flexible group-sequential approach was adopted. The general family of alpha spending function based on the rho-family with rho=2.5 at overall type I error of 0.025 (1-sided) was employed; Test type: Superiority or Other; p < 0.001, Weighted z-test — The two treatment groups were compared using a weighted z-statistic based on rho-family of alpha spending function at information fraction of 81.9% at interim analysis analysis (rho=2.5) at 0.025 (1-sided) level. One-sided alpha at final was 0.0198

3. Secondary Outcome: Time to Recurrence of Depressive Symptoms Associated With Bipolar I Disorder
Description: Pali/Pali and Pali/Placebo were compared with each other with respect to time to recurrence of depressive symptoms. The criterias used for this analysis were similar to criterias used for primary analysis.
Time Frame: Date of randomization into the maintenance phase until the first occurrence of recurrence of depressive symptoms or discontinuation from the study, assessed over a period of 41 months.
Population: Intent-to-treat analysis set in MA period, which included participants who entered the maintenance phase and took at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Number analyzed (Participants) | 0 | 0 | 144 | 146 | 82
Days |  |  | 503.0 [203.0 to NA] — There were 18% of the participants in the Pali/Placebo group who reported recurrence of depressive symptoms. | 448.0 [170.0 to 750.0] | NA [651.0 to NA] — There were 12% of the participants in the Olan/Olan group who reported recurrence of depressive symptoms. Hence the 25% quartile of the time to recurrence of depressive symptoms was not observed.
Statistical Analysis 1: Comparison: Pali/Placebo vs Pali/Pali; Test type: Superiority or Other; Regression, Cox — Cox proportional hazards regression was performed with treatment (Pali/Placebo, Pali/Pali) as a factor. The 2 treatment groups were compared by means of a hazard ratio (Pali/Placebo: Pali/Pali); The percent of participants who reported recurrence of depressive symptoms was: 18% Pali/Placebo, 24% Pali/Pali; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.53 to 1.46] — Hazard ratio was estimated with Pali/Placebo in the numerator and Pali/Pali in the denominator

4. Other Pre Specified Outcome: Young Mania Rating Scale (YMRS): Change From Baseline
Description: This is method by which condition of patient suffering with mania is checked. In this scale patient's condition is assessed using 11 items. A severity rating is assigned to each of 11 items based on the how subject feels of his or her condition and the physicians observation of patients behavior. The range of the scale is 0 to 60. A higher score indicates a more severe condition. Change from baseline (Day 105) in the double-blind maintenance phase to the last postbaseline assessment.
Time Frame: From 1st randomization into acute phase to end of acute/continuation phase (ie, up to 15 weeks after 1st randomization), or from randomization into maintenance (MA) phase to the end of MA phase (ie, up to 175 weeks (or 41 months) after 2nd randomization).
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Number analyzed (Participants) | 602 | 145 | 143 | 144 | 81
Scores on the scale | -19.2 (11.23) | -19.3 (10.25) | 9.0 (11.78) | 4.2 (9.33) | 1.3 (6.26)
Statistical Analysis 1: Comparison: Pali/Placebo vs Pali/Pali; Change from Baseline (Maintenance Phase) to Endpoint (Maintenance Phase); Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment group (Pali/Pali, Pali/Placebo) and country as factors with baseline value as covariate; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-6.92 to -1.98]

5. Other Pre Specified Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS consists of 10 items covering all the important complaints which patient with depression have (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Item is scored from 0 (normal) to 6 (severe). Total score (0 to 60) is calculated by adding the scores of all 10 items. A higher score represents a more severe condition. Negative Change in Score Indicates Improvement.
Time Frame: as for outcome 4
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Number analyzed (Participants) | 597 | 144 | 143 | 144 | 81
Scores on the scale | -2.7 (8.21) | -2.7 (7.82) | 6.0 (9.16) | 6.1 (10.10) | 2.5 (7.10)
Statistical Analysis 1: Comparison: Pali/Placebo vs Pali/Pali; Change from Baseline (Maintenance Phase) to Endpoint (Maintenance Phase); Test type: Superiority or Other; p = 0.763, ANCOVA; ANCOVA Model with treatment (Pali/Pali, Pali/Placebo) and country as factors with baseline value as covariate; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.87 to 2.55]

6. Other Pre Specified Outcome: Global Assessment of Functioning (GAF): Change From Baseline
Description: This scale is used when the clinical progress of a subject needs to be assessed in global terms, using a single measure. The GAF scale is rated with respect to psychological, social, and occupational functioning at the time of the assessment only. A higher score indicates a better functioning, with an overall range from 1 to 100. Positive Change in Score Indicates Improvement.
Time Frame: as for outcome 4
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Scores on the scale
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Number analyzed (Participants) | 575 | 137 | 131 | 135 | 77
Scores on the scale | 19.6 (17.38) | 20.8 (18.26) | -15.2 (20.93) | -8.9 (17.75) | -4.2 (13.98)
Statistical Analysis 1: Comparison: Pali/Placebo vs Pali/Pali; Change from Baseline (Maintenance Phase) to Endpoint (Maintenance Phase); Test type: Superiority or Other; p = 0.010, ANCOVA; ANCOVA Model with treatment (Pali/Pali, Pali/Placebo) and country as factors with baseline value as covariate; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [1.40 to 10.09]

7. Other Pre Specified Outcome: Clinical Global Impression - Bipolar Disorder - Severity of Illness (CGI-BP-S): Change From Baseline
Description: The CGI-BP-S rating scale is used to rate the severity of bipolar disorder, including both depressed and manic components, on a 7-point scale ranging from 1 (not ill) to 7 (very severely ill). This scale permits a global evaluation of the subject's bipolar condition at a given time. Negative Change in Score Indicates Improvement.
Time Frame: as for outcome 4
Population: Intent-to-Treat
Measure: Median (Full Range); unit: Scores on the scale
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Number analyzed (Participants) | 601 | 145 | 143 | 144 | 81
Scores on the scale | -2 [-6 to 2] | -3 [-5 to 2] | 2 [-1 to 6] | 0 [-2 to 5] | 0 [-1 to 4]
Statistical Analysis 1: Comparison: Pali/Placebo vs Pali/Pali; Change from Baseline (Maintenance Phase) to Endpoint (Maintenance Phase); Test type: Superiority or Other; p = 0.007, ANCOVA; ANCOVA Model on ranks with treatment (Pali/Pali, Pali/Placebo) and country as factors with baseline value as covariate

ADVERSE EVENTS:
Arm/Group | Paliperidone ER | Olanzapine | Pali/Placebo | Pali/Pali | Olan/Olan
Serious Adverse Events (participants affected / at risk) | 42/614 | 10/148 | 33/147 | 16/149 | 8/83
Other Adverse Events (participants affected / at risk) | 351/614 | 79/148 | 38/147 | 38/149 | 26/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=614) | Olanzapine (N=148) | Pali/Placebo (N=147) | Pali/Pali (N=149) | Olan/Olan (N=83)
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Hypoxic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Anger (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Catatonia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 4 | 1 | 8 | 4 | 1
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hypomania (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Mania (Psychiatric disorders) | 10 | 6 | 22 | 3 | 4
Pressure of speech (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Self-injurious ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 6 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Tachyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Breast operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Mastectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Nasal operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=614) | Olanzapine (N=148) | Pali/Placebo (N=147) | Pali/Pali (N=149) | Olan/Olan (N=83)
Dry mouth (Gastrointestinal disorders) | 28 | 14 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 33 | 2 | 2 | 1 | 0
Weight decreased (Investigations) | 7 | 0 | 9 | 4 | 1
Weight increased (Investigations) | 51 | 18 | 10 | 12 | 7
Increased appetite (Metabolism and nutrition disorders) | 23 | 13 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 83 | 11 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 41 | 4 | 1 | 4 | 0
Extrapyramidal disorder (Nervous system disorders) | 54 | 4 | 1 | 2 | 1
Headache (Nervous system disorders) | 78 | 14 | 7 | 4 | 7
Sedation (Nervous system disorders) | 38 | 25 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 76 | 23 | 0 | 5 | 1
Tremor (Nervous system disorders) | 34 | 4 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 83 | 15 | 14 | 13 | 7

LIMITATIONS AND CAVEATS:
The study employed a randomized withdrawal design, and as such, was enriched for responders to the study drug. Thus, the long-term efficacy demonstrated cannot be extrapolated to a population of patients without prior exposure to paliperidone ER.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days